CLINICAL TRIAL: NCT01028313
Title: A Phase II Study of Panobinostat (LBH589) as Second-Line Therapy in Patients With Chronic Graft-Versus-Host Disease
Brief Title: A Study of Panobinostat (LBH589) as Second-Line Therapy in Patients With Chronic Graft-Versus-Host Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision was made to not move forward with the study. No participants were enrolled or treated.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Daniel Couriel, MD, SCRI Oncology Research Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BMT 02
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Graft-Versus-Host Disease
Keywords: Chronic Graft-Versus-Host Disease; GVHD; LBH589; Panobinostat
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Panobinostat; Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Systemic Therapy
  Interventions: Drug: LBH589; Drug: Methylprednisolone

INTERVENTIONS:
Drug: LBH589 — 20 mg PO three times weekly
  Other Names: Panobinostat
Drug: Methylprednisolone — 1 mg/kg/day PO continuously
  Other Names: Medrol, Depo-Medrol

SUMMARY:
There is a clear need for effective, steroid-sparing agents for the management of chronic graft-versus-host disease (GVHD). Thus, agents like Histone deacetylase (HDAC) inhibitors, with the potential of decreasing pro-inflammatory events leading to GVHD without affecting graft-versus-leukemia (GVL), may have a central role in the prevention and treatment of GVHD.

This study will look at the efficacy of panobinostat (LBH589), an HDAC inhibitor, in the treatment of patients with chronic GVHD who have failed corticosteroids. In this group of patients, effective steroid-sparing options are limited and are usually associated with profound immunosuppression and decreased GVL effect.

DETAILED DESCRIPTION:
Chronic GVHD is an autoimmune, inflammatory disorder that occurs in the majority of patients who experience acute GVHD. Long-term corticosteroids are still standard therapy for chronic GVHD. Corticosteroids are associated with high morbidity and non-relapse mortality. In addition, corticosteroids are broadly immunosuppressive and can also decrease the GVL effect and increase the incidence of relapse. There is a clear need for effective, steroid-sparing agents for the management of chronic GVHD. Thus, agents like HDAC inhibitors, with the potential of decreasing pro-inflammatory events leading to GVHD without affecting GVL, may have a central role in the prevention and treatment of GVHD.

This study will look at the efficacy of panobinostat (LBH589), an HDAC inhibitor, in the treatment of patients with chronic GVHD who have failed corticosteroids. In this group of patients, effective steroid-sparing options are limited and are usually associated with profound immunosuppression and decreased GVL effect.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic GvHD following allogeneic HSCT of any source (bone marrow, peripheral blood, or cord blood stem cells), from any donor type (related, unrelated, or mismatched) and with any type of malignancy. Chronic GvHD will be defined according to NIH Consensus Criteria.
2. Patients must have had inadequate response to treatment with steroids and calcineurin inhibitors. Patients must have been treated with an initial dose of at least 1 mg/kg/day of methylprednisolone (MP) or equivalent in combination with tacrolimus or cyclosporine and must fulfill the definition of steroid refractoriness or resistance. Steroid refractoriness or resistance will be defined as:

   1. Lack of any response after 1 month of treatment with MP, including 15 days of at least 0.5 mg/kg/day.
   2. Worsening of existing GvHD or new organ involvement at any time following one week of initiation of MP at 1 mg/kg/day.
   3. Reflare or worsening of GvHD at any time during steroid taper.
   4. Patients should not have received any drug or treatment for chronic GvHD other than steroids and calcineurin inhibitors (i.e., cyclosporine or tacrolimus).
3. Patient must not have evidence of primary disease relapse.
4. An ECOG (Eastern Cooperative Oncology Group) performance status of ≤2
5. Baseline MUGA or ECHO must demonstrate left ventricular ejection fraction (LVEF) ≥40%.
6. No uncontrolled arrhythmias or symptoms of heart disease.
7. FEV1, FVC, and DLCO ≥40%.
8. Laboratory values as follows:

   * white blood cell ≥2500/mm³;
   * absolute neutrophil count (ANC) ≥1,000/mm³;
   * hemoglobin ≥9.5 g%;
   * platelets ≥50,000/mm³;
   * total bilirubin <3 x upper limits of normal;
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × the institutional upper limit of normal (ULN);
   * creatinine <1.5 × ULN or creatinine clearance ≥ 50 ml/min;
   * serum potassium ≥ LLN;
   * serum sodium ≥ LLN;
   * serum calcium WNL;
   * serum phosphorus WNL;
   * serum magnesium WNL;
9. Patients with elevated alkaline phosphatase due to bone metastasis may be enrolled.
10. TSH and free T4 within normal limits (clinically euthyroid patients are permitted to receive thyroid supplements to treat underlying hypothyroidism).
11. Age ≥ 18 years, male or female.
12. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer.
2. Patients who will need valproic acid for any medical condition during the study or ≤5 days prior to first panobinostat treatment.
3. Use of prior immunosuppressants other than steroids and calcineurin inhibitors(i.e. cyclosporine or tacrolimus).
4. Chronic active hepatitis or cirrhosis.
5. Impaired cardiac function including any of the following:

   * Patients with congenital long QT syndrome;
   * Patients with history or presence of sustained ventricular tachyarrhythmias;
   * Patients with any history of ventricular fibrillation or Torsades de Pointes;
   * Patients with bradycardia defined as HR <50 bpm. Patients with pacemakers are eligible if HR ≥50 bpm.
   * Patients with myocardial infarction or unstable angina ≤6 months prior to starting study drug;
   * Right bundle branch block plus left anterior hemiblock (bifasicular block);
   * Screening ECG with QTc >450 msec;
   * Congestive heart failure (CHF) > New York Heart Association (NYHA) Class II (see Appendix D).
6. Concomitant use of drugs with a risk of causing Torsades de Pointes (see Appendix A).
7. Other concurrent severe and/or uncontrolled medical conditions.
8. Any condition that impairs patient's ability to swallow whole pills or gastrointestinal (GI) tract disease that involves an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To assess the response rate to panobinostat of patients with cGvHD inadequately treated with steroids and calcineurin inhibitors. | 30 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of panobinostat in patients with cGvHD. | 30 months
To assess the steroid-sparing capacity of panobinostat (as proportion of patients able to discontinue steroids while receiving, or following therapy with, panobinostat). | 30 months
To assess changes in quality of life (QOL) after treatment with panobinostat. | 30 months
To analyze survival at 6 and 12 months after initiation of panobinostat. | 30 months
To evaluate the relapse rate of the underlying malignancy as well as the occurrence of second malignancies at 6 and 12 months after initiation of panobinostat. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Couriel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States